CLINICAL TRIAL: NCT05875766
Title: Evaluation of Osteopathic Care After Rupture of the Antero-external Cruciate Ligament of the Knee
Brief Title: Evaluation of Osteopathic Care After Rupture of the Antero-external Cruciate Ligament of the Knee (DIDT OSTEO)
Acronym: DIDT OSTEO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ramsay Générale de Santé (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-A00450-43
Record Dates: First submitted 2023-05-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Cruciate Ligament Rupture; Knee Ligament Injury; Osteopathia
MeSH Terms: conditions — Bone Diseases | interventions — Osteopathic Physicians; Physical Therapy Modalities

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient with osteopathy session (Experimental): Patients after their DIDT surgery have 4 osteopathy sessions in addition to physiotherapy
  Interventions: Other: Osteopathy; Other: Physiotherapy
- Patient without osteopathy session (Placebo Comparator): Patients after their DIDT surgery have only physiotherapy
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Osteopathy — 4 sessions of osteopathy after DIDT surgery
  Arms: Patient with osteopathy session
Other: Physiotherapy — Physiotherapy after DIDT surgery (reference treatment)

SUMMARY:
The antero-external cruciate ligament (ACL) is the ligament located inside the knee, which allows the rotation of the knee by stabilizing the femur and the tibia. Rupture of the ACL is common during the practice of certain so-called "pivot" sports, whether contact or not. It is manifested by acute pain or instability of the knee, following a crack during a twist and/or a blockage of the joint. The diagnosis will be confirmed by a clinical examination and X-rays to eliminate any fracture or tearing and by MRI to visualize the ligament rupture and the associated lesions, in particular a lesion of the meniscus.

Treatment is required because the ruptured ligament does not heal on its own and the rupture of the ligament may eventually promote the appearance of osteoarthritis. Two types of treatment can be considered, rehabilitation or surgery, depending on the patient's age and motivation to resume sports. There are several surgical techniques, the most common is to reconstruct the ruptured ligament by arthroscopy using a graft taken from the tendons of the Internal Rectus and Demi muscles tendinous (DIDT). Rehabilitation by physiotherapy is often started preoperatively and immediately after the operation, as soon as you wake up, to find a functional and painless knee. Functional recovery often depends on patient motivation.

The main objective is to show that osteopathic care in addition to physiotherapy rehabilitation improves knee functionality in patients 6 months after reconstruction of the ACL by DIDT.

ELIGIBILITY:
Inclusion Criteria:

* Patient, male or female, aged 18 to 35 inclusive
* Patient with a BMI between 18.5 and 30 kg/m² (limits included).
* Patient presenting with a total rupture of the unilateral anterior cruciate ligament (ACL).
* Candidate patient for reconstruction of the ACL with the DIDT method.
* Affiliated patient or beneficiary of a social security scheme.
* Patient having been informed and having given their free consent, enlightened and written.

Exclusion Criteria:

* Patient with damage to another structure of the knee, other than meniscal lesions.
* Patient with a contraindication to osteopathic intervention.
* Patient for whom a method other than DIDT has been proposed.
* Patient with iterative rupture of the ACL.
* Patient having undergone ligamentoplasty of the contralateral knee
* Patient participating in another research.
* Patient in period of exclusion from another research still in progress at the time of inclusion.
* Protected patient: adult under guardianship, curatorship or other legal protection, deprived of liberty by judicial or administrative decision.
* Pregnant, breastfeeding or parturient women.
* Patient hospitalized without consent.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 94 (Estimated)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-04-07 (Estimated); Study Completion 2024-12-07 (Estimated)

PRIMARY OUTCOMES:
assess the functionality of the knee | 6 months
  Using International Knee Documentation Committee Subjective Knee Form (IKDC) measured 6 months postoperative and referring to the last weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital privé Jean Mermoz, Lyon, France